CLINICAL TRIAL: NCT04382365
Title: Use of an Internet-Based Insomnia Intervention to Prevent Cognitive Decline in Adults With Mild Cognitive Impairment
Acronym: SHUTi OASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Meghan Mattos, Assistant Professor of Nursing, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-HSR #20990
Record Dates: First submitted 2020-05-04; First posted 2020-05-11 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Mild Cognitive Impairment; Cognitive Impairment; Insomnia
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-Based Insomnia Intervention (Other): 2 weeks of online sleep diaries. Participants will also wear an Actiwatch at night, which records measurements of movements of a limb, providing an estimation of sleep duration, sleep pattern and disturbed sleep.
  9 week interveition period, subjects complete the internet based CBT-I program, consisting of six Cores (Getting Ready, Sleep Scheduling, Sleep Practices, Thinking Differently, Sleep Hygiene, and Moving On).Each Core takes approximately 45-60 minutes to review online, and most participants spend an additional 30-45 minutes per week on recommended exercises.
  Participant will then be instructed to complete a post-Assessment, consisting of one online questionnaire and two weeks of Daily Sleep Diaries. The Actiwatch is worn as before during this two week period.
  Interventions: Other: Sleep Health Using the Internet for Older Adult Sufferers of Insomnia and Sleeplessness

INTERVENTIONS:
Other: Sleep Health Using the Internet for Older Adult Sufferers of Insomnia and Sleeplessness — Cognitive-Behavioral Treatment for insomnia (CBT-I) is a non-pharmacological intervention that is effective in treating insomnia in older adults, even when present with comorbid medical and psychological conditions.25 CBT-I focuses on the maladaptive behaviors and dysfunctional thoughts that perpetuate sleep problems, and typically consists of five primary treatment components: sleep restriction, stimulus control, cognitive restructuring, sleep hygiene, and relapse prevention.

SUMMARY:
The purpose of the study is to determine feasibility of an online program providing cognitive behavioral therapy for insomnia in adults with cognitive impairment.

The study involves the use an Internet program (website) for 9 weeks. There are two required study visits in the home or in a UVA clinic. Participants will complete online questionnaires and sleep diaries twice during a 4-month period. Participants will also wear a sleep watch for two weeks before and after using the website.

DETAILED DESCRIPTION:
Mild cognitive impairment in older adults. Mild Cognitive Impairment (MCI) is recognized as an early stage cognitive disorder, a condition where patients live independently and are able to still perform many instrumental activities of daily living.1,2 Individuals with MCI typically present with subtle cognitive changes that can worsen over time.3,4 MCI prevalence is estimated to be as high as 19% among older adults in the US,3,5 with 10-13% progressing to dementia, such as Alzheimer's disease (AD), every year.6-8 With no known cure for MCI, current treatments focus on the maintenance of cognitive function, management of behavioral symptoms, and slowing or delaying the symptoms of disease.9 Characteristics of sleep in MCI and AD. Recent research concludes that individuals with cognitive impairment experience more disruptive sleep and sleep disorders than those without cognitive concerns.10-12 Older adults also more likely to have MCI, and other age-related sleep changes include a decrease in total sleep duration, decreased sleep efficiency, increased sleep fragmentation, increased sleep onset latency, and decreased slow wave and rapid eye movement (REM) sleep. In a review examining the effect of poor sleep on cognitive outcomes, poor sleep was identified as a risk factor for cognitive decline and AD.10 Recent research seeks to understand the mechanisms underlying this relationship using neuroimaging as well as sleep and cognitive functioning data. Although exact mechanisms underlying this relationship are not yet known, and possibly interactive, healthy sleep promotes maintenance of brain health, and may delay symptoms of AD and other dementias.10 Insomnia in older adults. Insomnia affects up to 25% of older adults. It is characterized by difficulty falling asleep and/or maintaining sleep as well as impaired functioning during waking hours.13 Individuals with insomnia have decreased work productivity, more accidents, more hospitalizations, and overall greater healthcare costs compared to their healthy counterparts.14,15 Insomnia symptoms can also affect significant others and caregivers. Specifically, nighttime activities can disrupt partners' sleep, which may impact the ability for him or her to function normally and provide care, as insomnia has been associated with decrease in measures of attention.16,17 Although everyone is at risk for developing insomnia, there are certain factors that increase one's risk. For example, predisposing factors include older age, female gender, and a positive family history of sleep disorders.18 The most common precipitating factors are psychological stress and major life changes. Factors known to perpetuate insomnia are typically behavioral and cognitive reactions, which are learned responses to sleep problems (e.g., daytime napping).

Treatment of insomnia. Treatment is recommended in two forms: pharmacological and behavioral-based interventions. Most commonly, sleep disturbances are treated with medication.19 Although pharmacological interventions can be effective in the short-term, they do not treat underlying predisposing, precipitating, and/or perpetuating factors of insomnia. Older adults experience pharmacokinetic and pharmacodynamic changes associated with aging;20 are more susceptible to consequences of potentially inappropriate medications;21 and are most likely to experience negative side-effects of polypharmacy.22 Age-related issues are especially concerning when using traditional benzodiazepines and non-benzodiazepine receptor agonist sleep aids such as zolpidem, eszopiclone, and zaleplon. Use of traditional sleep aids in older adults has been associated with serious adverse events (e.g., cognitive impairment, falls).23,24 Despite evidence regarding adverse consequences, pharmacological treatment of insomnia remains the most common treatment for insomnia.

Non-pharmacological treatment of insomnia. Cognitive-Behavioral Treatment for insomnia (CBT-I) is a non-pharmacological intervention that is effective in treating insomnia in older adults, even when present with comorbid medical and psychological conditions.25 CBT-I focuses on the maladaptive behaviors and dysfunctional thoughts that perpetuate sleep problems, and typically consists of five primary treatment components: sleep restriction, stimulus control, cognitive restructuring, sleep hygiene, and relapse prevention.26,27 Although there are effective treatments for insomnia, less than 15% of all adults with chronic insomnia are estimated to get any treatment for insomnia.28 Even for those seeking CBT-I, access is extremely limited due to the small number of clinicians trained in behavioral insomnia treatment.29 Internet CBT-I. The Internet has the potential to overcome barriers related to obtaining face-to-face CBT-I. Older adults have historically had limited Internet access, but this is changing dramatically. In 2000, only 14% of adults over the age of 64 used the Internet.30 In 2017, 66% of adults over 65 years of age and 87% age 50-64, reported Internet access.30 Almost 50% of older adults describe the Internet as ''quite a bit'' to ''extremely'' helpful to find new knowledge about their disease, treatment options, and drug therapy.59 Older adults are also more likely to use technology when presented with the potential benefits.57 Internet-delivered interventions for older adults have also been shown to be feasible and effective. For example, Internet-delivered interventions for dementia caregivers improved caregiver confidence, depression, and self-efficacy.31 The CBT-I internet intervention, Sleep Healthy Using Internet (SHUTi) for Older Adult Sufferers of Insomnia and Sleeplessness (OASIS), was developed for adults over age 55.

Sleep diaries and actigraphy. Sleep diaries are often used both as a behavioral tool during CBT-I as well as a way to determine the effect of CBT-I on sleep. For the latter, sleep diaries are kept by the patient both prior to and following the intervention and the patient reports on various sleep factors each night. From this self-reported data, sleep variables can be calculated, such as sleep onset latency (SOL), wakefulness after initial sleep onset (WASO), total sleep time (TST), total time spent in bed (TIB), sleep efficiency (SE), and sleep quality.32 This data can also be collected passively through the use of actigraphy. Actigraphy is an objective, non-invasive, and minimally burdensome approach to continuously measure gross motor activity and provide wake/sleep timing. Although actigraphy is considered less reliable in patients with insomnia compared to polysomnography (PSG),33 actigraphy provides the opportunity to collect multiple nights at little to no extra burden to participants. There is also a strong correlation between sleep diaries and actigraphy. Most notably, Chambers34 found a substantial within-participant correlation (r = .80) between actigraph and sleep diaries, and, we plan to use actigraphy for similar within-participant analyses examining sleep variability and patterns.

The proposed research focuses on individuals with Mild Cognitive Impairment and insomnia, positing that improved sleep will moderate further cognitive decline. Before undertaking large-scale interventions to determine efficacy of SHUTi OASIS in this population and long-term cognitive outcomes of improved sleep, there must be preliminary work to determine feasibility of delivering the intervention to older adults with MCI and insomnia. To better understand sleep patterns of individuals with MCI and insomnia, actigraphy data will be collected and analyzed to identify within-participant sleep patterns.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older

  * ability to read and speak English
  * US resident
  * MCI diagnosis or scores within acceptable range on R-BANS assessment.
  * regular access to Internet and Email
  * willingness to use Internet and Email
  * ability to use a computer
  * no more than 6.5 hours of sleep per night
  * the sleep disturbance (or associated daytime fatigue) must cause significant distress or impairment in social, occupational, or other areas of functioning over past 3 months
  * sleep onset latency > 30 minutes at least 3x/week for past three months; OR wake after sleep onset >30 minutes at least 3x/week for past three months

Participants on stable (defined as no change in the past 3 months) medication regimens will be eligible including sleep medications, unless the medication is known to cause insomnia (e.g., steroids).

Exclusion Criteria:

* bedtime outside of 8pm-2am and arise times outside of 4-10am

  * current psychological treatment for insomnia
  * initiation of psychological or psychiatric treatment within past 3 months
  * current severe/very severe depression from QIDS-C16
  * current moderate/high risk suicide or substance use disorder in 12 months from MINI
  * other untreated sleep disorders (e.g., obstructive sleep apnea, restless legs syndrome)
  * current diagnosis of Huntington's or Parkinson's disease
  * current treatment for hyperthyroidism
  * currently undergoing chemotherapy
  * presence of asthma or respiratory concerns with night treatment
  * chronic pain treated with opioids
  * epilepsy
  * inability to provide informed consent
  * Not concurrently enrolled in any other intervention or educational study targeting sleep.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Increase in Sleep Duration | Baseline
  Patient generated data on sleep through questionnaires
Increase in Sleep Duration | 11 weeks
  Patient generated data on sleep through questionnaires
Impact on Psychological Distress | Baseline
  Patient generated data on sleep through questionnaires
Impact on Psychological Distress | 11 weeks
  Patient generated data on sleep through questionnaires
Impact on Overall Health | Baseline
  Patient generated data on sleep through questionnaires
Impact on Overall Health | 11 weeks
  Patient generated data on sleep through questionnaires
Impact on Sleep Pattern | Baseline
  Data obtained through wrist actigraphy.
Impact on Sleep Pattern | 11 weeks
  Data obtained through wrist actigraphy.

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Virginia, Charlottesville, Virginia, United States